CLINICAL TRIAL: NCT01348867
Title: A Randomised Study to Evaluate the Effectiveness of a Treat-to-target Clinic Led by a Nurse Consultant in Managing Patients With Type 2 Diabetes in Hong Kong
Brief Title: Effectiveness of a Treat-to-target Clinic Led by a Nurse Consultants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asia Diabetes Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CRE-2009-394
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2011-05

CONDITIONS: Diabetes
Keywords: Diabetes; Structured Care
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): These 120 controls will undergo a comprehensive assessment at baseline then again at 12 months, which is similar to the intervention group. However, in between these 2 time points the 'control' patients will receive usual care and hence will not be monitored under the structured care protocol by a diabetes nurse consultant led team.
- Structured Care (Experimental): 120 patients will be randomised to the structured care group, and these patients will receive repeated follow-ups and contact with the structured care team in between the two comprehensive assessments at week 0 and week 52.
  Patients will be seen by Diabetes Nurse Consultant at week 0, 6, 12, 24 38 during the year. At each visit, clinical and laboratory measurements will be performed; treatment compliance and self care will be assessed and medications will be adjusted to optimise metabolic and cardiovascular risk factors control.
  Patients will be seen by the doctors in their clinic follow up at week 0, 24 and 52.
  Technical service assistance will telephone patient at week 18, 30 and 44 to reinforce patient to take medications, attend clinical follow up.
  Interventions: Other: Structured care led by a nurse consultant

INTERVENTIONS:
Other: Structured care led by a nurse consultant — For the intervention group, patients will be followed up according to the following protocol. The structured care team consists of:
  i) Diabetes Nurse Consultant to reinforce compliance; educate patients on insulin injection techniques and reinforce self-care including self blood glucose monitoring and lifestyle interventions, titration of medication.
  ii) Technical Service Assistance to remind patients to take medications and/or give insulin injection, monitor blood glucose as prescribed, attend their next clinic appointment, encourage patients to report all side effects, self initiated change in regimen or concerns to diabetes nurse consultant and/or their doctors at the next follow up visit.
  Arms: Structured Care

SUMMARY:
The investigators hypothesize a diabetes nurse consultant led team with particular emphasis on compliance and attainment of treatment targets in Type 2 diabetic patients will achieve metabolic control, improve clinical outcomes and levels of self efficacy compared to usual clinic-based care.

DETAILED DESCRIPTION:
Diabetes patients consume over 10% of health care costs in most developed countries. Over 80% of these resources are used to treat diabetic complications and late stage diseases. In Hong Kong, the prevalence of diabetes was reported to be 10%. Over 30% of patients admitted to the medical wards in Hong Kong's public hospitals have diabetes, mainly due to cardiovascular and renal complications. The number of patients receiving renal replacement therapy has increased by 50% in the last 5 years but the number of patients with end stage renal disease due to diabetes has doubled. Between 10% and 15% of patients attending medical clinics in local public hospitals either receive insulin or anti-diabetic drugs. Local published data show that 3-10% of diabetic patients died or developed clinical endpoints yearly.

There are now overwhelming evidence supporting the beneficial effects of optimal control of cardiovascular risk factors on clinical outcomes in diabetic patients. However, there are few studies to examine the most effective way to translate these evidence collected in closely monitored clinical trials situations into daily clinical practice. Against this background, the investigators hypothesize that disease management using a team approach to implement a structured care model in daily clinical practice will improve the clinical outcomes in high risk Type 2 diabetic patients compared to usual clinic-based care with no specific built in protocol and/or monitoring mechanism to ensure its effective implementation. The nurse consultant led clinics will use a structured protocol with particular emphasis on periodic monitoring, treating to target and reinforcing patient adherence.

In light of the size of diabetes epidemic, the constraints of finite resources and the need for equity, the investigators propose the results from this randomized study will provide information to health care policy makers regarding the effectiveness of diabetes nurse consultant led clinics in managing diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients
* Aged between 18 and 75 years (inclusive)
* HbA1c >8%
* Chinese in ethnicity
* patients under the care of clinicians who aimed the treatment targets of their patients as HbA1c <7%, BP <130/80 mmHg, and LDL-C <2.6 mmol/L

Exclusion Criteria:

* patients with clinically unstable psychiatric illnesses
* patients with terminal malignancy or other life-threatening diseases with less than 3-month expected survival
* patients who speak non-Cantonese dialect or a different language or have conditions that prevent effective face-to-face or telephone communications eg. Patients who are deaf or mute
* patients who live in nursing home with supervised treatment
* patients who are not available via telephone contact

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To assess the effectiveness of the nurse consultant led clinic in improving glycemic parameters in patients with type 2 diabetes | 12 months
  Metabolic parameters such as HbA1c, blood pressure, lipid profile, body mass index (BMI) etc, will measured at specific time points throughout the study

SECONDARY OUTCOMES:
To assess the any changes in diabetic knowledge, behaviours and level self-efficacy of the participants as compared to the control patients | 12 months
  The cognitive psychosocial-behavior assessment will include using the Summary of Diabetes Self- Care Activities (SDSCA), Diabetes Empowerment Scale (DES), Depression Anxiety Stress Scale-21 (DASS21), General Health Questionnaire (GHQ12).
A comparison of the patients' utility of healthcare services | 12 months
  The number of hospital admissions, total number of days stay in hospital, number of attendances at Accident and Emergency department will be explored and compared for all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Wong, Principal Investigator — Prince of Wales Hospital, Shatin, Hong Kong
Locations (1):
- Diabetes & Endocrine Centre, Prince of Wales Hospital, Shatin, New Territories, Hong Kong

REFERENCES:
- See also: Works of the Asia Diabetes Foundation — http://www.adf.org.hk